CLINICAL TRIAL: NCT03862794
Title: A Randomized Controlled Trial of Behaviourally Informed Feedback Letters Sent by the Chief Medical Officer on the Amount of Antibiotics and the Percentage of Broad Spectrum Antibiotics Prescribed in Primary Care
Brief Title: CMO Letter to Reduce Unnecessary Antibiotic Prescribing and Broad Spectrum Prescribing Winter 2018-9
Acronym: CMO2018-9
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R&D 193
Record Dates: First submitted 2019-02-27; First posted 2019-03-05 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2018-12

CONDITIONS: Prescribing, Off-Label

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- high total and high broad spectrum prescribing letter (Experimental): social norm feedback letter with bar chart GPs who prescribe more than 1.161 Antibacterial Items/ STAR-PU and more than 10% broad spectrum receive a letter that has specific information about the percentile they are on for broad spectrum prescribing and a bar chart representing their broad spectrum prescribing compared to the average
  Interventions: Behavioral: new social norm feedback letter with bar chart
- high total and high broad spectrum prescribing control (Active Comparator): standard social norm feedback letter GPs who prescribe more than 1.161 Antibacterial Items/ STAR-PU and more than 10% broad spectrum receive the standard practice overall prescribing letter as a control
  Interventions: Behavioral: standard social norm feedback letter
- high total prescribing only intervention letter (Experimental): social norm feedback letter with bar chart GPs who prescribe more than 1.161 Antibacterial Items/ STAR-PU and less than 10% broad spectrum receive a letter that has specific information about the percentile they are on for overall prescribing and a bar chart representing their overall prescribing compared to the average
  Interventions: Behavioral: new social norm feedback letter with bar chart
- high total prescribing control letter (Active Comparator): standard social norm feedback letter GPs who prescribe more than 1.161 Antibacterial Items/ STAR-PU and less than 10% broad spectrum receive the standard practice overall prescribing letter as a control
  Interventions: Behavioral: standard social norm feedback letter
- moderate total prescribing and high broad spectrum letter (Experimental): social norm feedback letter with bar chart GPs who prescribe more than 0.965 but less than 1.161 Antibacterial Items/ STAR-PU and more than 10% broad spectrum will receive a letter that has specific information about the percentile they are on for broad spectrum prescribing and a bar chart representing their broad spectrum prescribing compared to the average
  Interventions: Behavioral: new social norm feedback letter with bar chart
- moderate total prescribing and high broad spectrum control (No Intervention): GPs who prescribe more than 0.965 but less than 1.161 Antibacterial Items/ STAR-PU and more than 10% broad spectrum receive no letter, which is standard practice, as a control.

INTERVENTIONS:
Behavioral: new social norm feedback letter with bar chart — letter with the percentile prescribing the practice is on and a bar chart, comparing prescribing to the national average
  Arms: high total and high broad spectrum prescribing letter; high total prescribing only intervention letter; moderate total prescribing and high broad spectrum letter
Behavioral: standard social norm feedback letter — social norm feedback letter used as standard practice, without specific information about the prescribing percentile
  Arms: high total and high broad spectrum prescribing control; high total prescribing control letter

SUMMARY:
This trial aims to reduce unnecessary prescription of antibiotics and broad spectrum antibiotics by general practitioners (GPs) in England. Unnecessary prescriptions are defined as those that do not improve patient health outcomes. The intervention is to send GPs a letter from the Chief Medical Officer (CMO) that gives feedback on their practice's prescribing levels. Specifically the sample was GPs whose practices whose prescribed more than 1.161 items per STAR-PU or whose practices prescribed more that .965 items per STAR-PU and greater than 10% broad spectrum items. The intervention groups received a letter telling them they are among the highest prescribers of either their total or broad spectrum antibiotics, with a graph showing their prescribing compared to average prescribing ("their peers"). The letter also contained a leaflet to help GPs discuss self-care advice with patients and some advice to use delayed prescriptions. The investigators hypothesize that the antibiotic prescribing rate in will be lower for the treatment group compared to the control group, following the receipt of the letter.

ELIGIBILITY:
Inclusion Criteria:

* GP practices that prescribed more than 1.161 Antibacterial Items/STAR-PU for the twelve months (June 2017 - May 2018)
* GP practices that prescribed more than 0.965 Antibacterial Items/STAR-PU and also more than 10% broad spectrum items for the twelve months (June 2017 - May 2018).

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7000 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
total antibiotic prescribing weighted by Specific Therapeutic group Age-sex Related Prescribing Unit (STAR-PU) in November for each GP practice | 1 month
  antibiotic prescribing weighted by Specific Therapeutic group Age-sex Related Prescribing Unit (STAR-PU)
total broad spectrum antibiotic prescribing weighted by STAR-PU in November for each GP practice | 1 month
  broad spectrum antibiotic prescribing weighted by Specific Therapeutic group Age-sex Related Prescribing Unit (STAR-PU)
percentage broad spectrum antibiotic prescribing in November for each GP practice | 1 month
  percentage broad spectrum antibiotic prescribing
total non-broad spectrum antibiotic prescribing weighted by STAR-PU in November for each GP practice | 1 month
  total overall antibiotic prescribing minus total broad spectrum antibiotic prescribing
total antibiotic prescribing weighted by STAR-PU in December for each GP practice | 2 months
  antibiotic prescribing weighted by Specific Therapeutic group Age-sex Related Prescribing Unit (STAR-PU)
total broad spectrum antibiotic prescribing weighted by STAR-PU in December for each GP practice | 2 months
percentage broad spectrum antibiotic prescribing in December for each GP practice | 2 months
total non-broad spectrum antibiotic prescribing weighted by STAR-PU in December for each GP practice | 2 months
total antibiotic prescribing in January weighted by STAR-PU for each GP practice | 3 months
total broad spectrum antibiotic prescribing weighted by STAR-PU in January for each GP practice | 3 months
percentage broad spectrum antibiotic prescribing in January for each GP practice | 3 months
total non-broad spectrum antibiotic prescribing weighted by STAR-PU in January for each GP practice | 3 months
total antibiotic prescribing weighted by STAR-PU in February for each GP practice | 4 months
total broad spectrum antibiotic prescribing weighted by STAR-PU in February for each GP practice | 4 months
percentage broad spectrum antibiotic prescribing in February for each GP practice | 4 months
total non-broad spectrum antibiotic prescribing weighted by STAR-PU in February for each GP practice | 4 months
total antibiotic prescribing weighted by STAR-PU in March for each GP practice | 5 months
total broad spectrum antibiotic prescribing weighted by STAR-PU in March for each GP practice | 5 months
percentage broad spectrum antibiotic prescribing in March for each GP practice | 5 months
total non-broad spectrum antibiotic prescribing weighted by STAR-PU in March for each GP practice | 5 months
total antibiotic prescribing weighted by STAR-PU in April for each GP practice | 6 months
total broad spectrum antibiotic prescribing weighted by STAR-PU in April for each GP practice | 6 months
percentage broad spectrum antibiotic prescribing in April for each GP practice | 6 months
total non-broad spectrum antibiotic prescribing weighted by STAR-PU in April for each GP practice | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Public Health England, London, United Kingdom

REFERENCES:
- [Derived] Gold N, Sallis A, Saei A, Arambepola R, Watson R, Bowen S, Franklin M, Chadborn T. Using text and charts to provide social norm feedback to general practices with high overall and high broad-spectrum antibiotic prescribing: a series of national randomised controlled trials. Trials. 2022 Jun 18;23(1):511. doi: 10.1186/s13063-022-06373-y. PMID 35717262